CLINICAL TRIAL: NCT01695304
Title: Pilot Intervention Trial of Ceramic Water Filters to Reduce the Burden of Cryptosporidium in Household Drinking Water in Rural Kenya.
Brief Title: Trial of Ceramic Water Filters to Reduce Cryptosporidium Infection in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCEZID-6369; CDCEID10A.1 (Other: Centers for Disease Control and Prevention); 2439 (Other: Kenya Medical Research Institute)
Record Dates: First submitted 2012-09-26; First posted 2012-09-27 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2015-09

CONDITIONS: Cryptosporidium; Diarrhea; Cryptosporidiosis; Communicable Diseases; Diarrheal Disease
Keywords: Cryptosporidiosis; Waterborne disease; Diarrheal disease; Ceramic water filters; infants; young children; drinking water; Kenya
MeSH Terms: conditions — Diarrhea; Cryptosporidiosis; Communicable Diseases; Waterborne Diseases

STUDY DESIGN:
Masking Description: This is an intervention trial of ceramic water filters, and as such cannot be masked. The intervention participants received the CWFs during the trial and the control group after the trial was over.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Arm (Experimental): Households with a child 4-10 months old will receive a Cera Maji ceramic water filter for treatment of drinking water.
  Interventions: Other: Ceramic water filter
- Control Arm (No Intervention): Households with a child 4-10 months old at initial entry into the study will not receive a ceramic water filter (control group). The study duration will be 6 months. All households in the control group will receive a Cera Maji ceramic water filter when the study ends.

INTERVENTIONS:
Other: Ceramic water filter — In total, 120 households with a child 4-10 months old will receive a Cera Maji ceramic water filter for treatment of drinking water at initial entry into the study (intervention group), and 120 households with a child 4-10 months old at initial entry into the study will not receive a ceramic water filter (control group). The study duration will be 6 months. All households in the control group will receive a Cera Maji ceramic water filter when the study ends.
  Other Names: Cera Maji ceramic water filter
  Arms: Intervention Arm

SUMMARY:
The aim of the study is to examine the efficacy of ceramic water filters to reduce the burden of waterborne diarrheal illness among infants in selected villages in Kenya. In Kenya very young children are given drinking water or water is used in reconstitution of their food. We hypothesize that ceramic water filters will remove Cryptosporidium from drinking water reducing infection in infants.

DETAILED DESCRIPTION:
Diarrhea is a major cause of illness among children in Africa. Cryptosporidium is a protozoan waterborne diarrheal pathogen resistant to chlorine. Ceramic filters are effective at improving drinking water quality, including removal of protozoa. In a recent preliminary analysis of >22,000 children <5 years enrolled in the Global Enterics Multi-Center Study (GEMS) case-control study of moderate-to-severe diarrhea, Cryptosporidium was identified as a leading cause of diarrhea in infants across all four participating African sites. This pilot is the first Cryptosporidium specific intervention trial of household ceramic water filters to reduce the burden of cryptosporidiosis acquired through drinking water in rural Kenya.

ELIGIBILITY:
Inclusion Criteria:

Children 4-10 months old living in selected villages in the Asembo Health and Demographic Surveillance System (HDSS) study area in Kenya whose primary caretakers consent on their behalf to be visited weekly for 6 months to carry out weekly illness surveillance, and have a follow up home visit one year after initial enrollment into the trial. The household in which the child resides must be a consenting participant in the HDSS. As the children included in the trial are infants, the child's primary caretaker will be invited to participate and be administered questionnaires. Random selection will be at the compound level. Only one household per compound will be eligible for selection.

Exclusion Criteria:

Children 4-10 months old whose households are not active consenting participants in the HDSS will not be eligible for inclusion. Only the subset of children 4-10 months old who are randomly selected in the sample will be eligible for participation.

-

Ages: 4 Months to 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 227 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Mintz, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Kemri/Cdc, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
No PII will be shared with any researcher. It is possible that researchers may request access to the clean de-identified data once closed out for all aspects of the work.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 120 | 120
Completed | 120 (2 deaths & 1 drop out in the intervention group, contributed some information over the 26 weeks) | 120 (3 deaths & 2 drop out in the intervention group, contributed some information over the 26 weeks)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Continuous [Median (Full Range); unit: months] | 7 [4 to 10] | 8 [4 to 10] | 7.5 [4 to 10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 62 | 128
  Male | 54 | 58 | 112
Race/Ethnicity, Customized [Number; unit: participants]
  Luo ethnic group | 120 | 120 | 240
Region of Enrollment [Number; unit: participants]
  Kenya | 120 | 120 | 240

OUTCOME MEASURES:

1. Primary Outcome: Longitudinal Diarrhea Prevalence
Description: The primary outcome measure is the longitudinal prevalence of diarrheal disease.
Time Frame: 6 months
Population: Incidence rate per 100 person-weeks of observation
Measure: Number; unit: Incidence rate per 100 person-weeks
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 115 | 112
Incidence rate per 100 person-weeks | 7.6 | 8.9

2. Primary Outcome: Health Facility Visits for Diarrheal Disease
Description: incidence rate of health facility visits for diarrheal disease per 100 person-week of observation
Time Frame: 6 months
Population: incidence rate of health facility visits for diarrheal disease per 100 person-week of observation
Measure: Number; unit: incidence rate per 100 person-weeks
Groups:
- Intervention Group: Intervention group who received ceramic water filters
- Control Group: Control Group who did not receive ceramic water filters (until after the trial ended)
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 115 | 112
incidence rate per 100 person-weeks | 1.2 | 2.2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 2/120 | 3/120
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120
Other Adverse Events (participants affected / at risk) | 0/120 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes